CLINICAL TRIAL: NCT04247139
Title: Effect of Traditionally and Commercially Prepared Kefir on Cholesterol Levels in Adult Males With Borderline High Cholesterol Levels
Brief Title: Kefir Cholesterol Lowering Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00087964
Record Dates: First submitted 2020-01-22; First posted 2020-01-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-01

CONDITIONS: Hypercholesterolemia
Keywords: high cholesterol, kefir
MeSH Terms: conditions — Hypercholesterolemia | interventions — Kefir

STUDY DESIGN:
Who Masked: Participant
Masking Description: Both types of kefir will be flavoured the same, and visually look the same.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Commercial Kefir (Experimental): Commercially produced kefir
  Interventions: Other: Kefir
- Traditional Kefir (Experimental): Traditionally grown kefir
  Interventions: Other: Kefir

INTERVENTIONS:
Other: Kefir — commercial versus traditional kefir

SUMMARY:
High cholesterol (a type of fat in humans blood) may be one factor that can lead to heart disease. If people have higher cholesterol, it is possible that kefir (a food similar to yogurt) may help to control blood cholesterol levels.

DETAILED DESCRIPTION:
New research shows that kefir (which contains bacteria also known as microbes), similar to yogurt, may improve health by lowering cholesterol levels. Much of this research however, focuses on traditional types of kefir, which differ significantly from commercially prepared kefir with regards to the types of microbes in each kefir. Additionally, there is a lack of research looking at how commercial kefir compares to traditional kefir in its ability to improve health. This has led to the consumer being confused about the health benefits they believe they are receiving, such as reduced weight gain, and improved cholesterol levels, when they purchase and consume commercial kefir. The researchers have produced a commercially usable kefir that has the health benefits of traditional grain fermented kefir. This was accomplished with only a small subset of microbes present in the traditional kefir, leading to a much easier product to commercialize and produce. Thus, this study aims to look at whether kefir, produced in the researchers laboratory and commercially available kefir, given to males for in two separate months, results in any cholesterol lowering effects. Successful completion of this project could potentially result in the development of a new commercial kefir with health benefits that are supported by scientific research and testing. In addition, if positive results are seen, a larger study will be carried out to ensure that results of the current study are consistent for the Canadian population.

ELIGIBILITY:
Inclusion Criteria:

1. Males, aged 18-65y
2. Moderately hypercholesterolemic adults: LDL-C between 3.2 and 4.9 mM, but otherwise healthy
3. No history of CVD, type 2 diabetes, monogenic dyslipidemia or use of medications for hyperlipidemia (including statins).
4. No dairy allergy

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male participants
Enrollment: 21 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Change in Blood Lipids following provision of each type of Kefir | 4 weeks
  Change in blood lipid panel (HDL, LDL, Total Cholesterol, Triglycerides) will be measured in blood samples.

SECONDARY OUTCOMES:
Fecal microbiota composition changes following the provision of each type Kefir | 4 weeks
  16SrRNA-sequencing and whole metagenome sequencing will performed to determine gut microbial community changes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No